CLINICAL TRIAL: NCT02859961
Title: A Phase 2b/3, Multicenter Study to Assess the Treatment Strategy of Using PRO 140 SC As Long-Acting Single-Agent Maintenance Therapy for 48 Weeks in Virologically Suppressed Subjects with CCR5-tropic HIV-1 Infection
Brief Title: Study of PRO 140 SC As Single Agent Maintenance Therapy in Virally Suppressed Subjects with CCR5-tropic HIV-1 Infection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CytoDyn, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO 140_CD03
Record Dates: First submitted 2016-07-13; First posted 2016-08-09 (Estimated); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: HIV
MeSH Terms: interventions — leronlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- PRO 140 SC 350 mg weekly injection (Group A) (Experimental): PRO 140 350 mg (175 mg/mL) SC injections per week
  Interventions: Drug: PRO 140 (350 mg)
- PRO 140 SC 525 mg weekly injections (Group B) (Experimental): PRO 140 525 mg (175 mg/mL) SC injections per week
  Interventions: Drug: PRO 140 (525 mg)
- PRO 140 SC 700 mg weekly injections (Group C) (Experimental): PRO 140 700 mg (175 mg/mL) SC injections per week
  Interventions: Drug: PRO 140 (700 mg)

INTERVENTIONS:
Drug: PRO 140 (350 mg) — PRO 140 350 mg (175 mg/mL) SC injection per week
  Other Names: Leronlimab
  Arms: PRO 140 SC 350 mg weekly injection (Group A)
Drug: PRO 140 (525 mg) — PRO 140 525 mg (175 mg/mL) SC injection per week
  Other Names: Leronlimab
  Arms: PRO 140 SC 525 mg weekly injections (Group B)
Drug: PRO 140 (700 mg) — PRO 140 700 mg (175 mg/mL) SC injection per week
  Other Names: Leronlimab
  Arms: PRO 140 SC 700 mg weekly injections (Group C)

SUMMARY:
This study is a Phase 2b/3, multi-center study designed to evaluate the efficacy, safety, and tolerability of the strategy of shifting clinically stable patients receiving suppressive combination antiretroviral therapy to PRO 140 monotherapy and maintaining viral suppression for 48 weeks following study entry.

Consenting patients will be shifted from combination antiretroviral regimen to weekly PRO 140 monotherapy for 48 weeks during the Treatment Phase with the one week overlap of existing retroviral regimen and PRO 140 at the beginning of the study treatment and also one week overlap at the end of the treatment in subjects who do not experience virologic failure.

DETAILED DESCRIPTION:
The primary objective is to assess the treatment strategy of using PRO 140 SC as long-acting, single-agent maintenance therapy for the chronic suppression of CCR5-tropic HIV-1 infection. In addition, the prognostic factors of therapeutic success of PRO 140 monotherapy will be evaluated.

The secondary objective of the trial is to assess the clinical efficacy, safety and tolerability parameters following substitution of combination antiretroviral therapy with weekly PRO 140 monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age ≥18 years
2. Receiving combination antiretroviral therapy for last 24 weeks
3. No change in ART within last 4 weeks prior to Screening Visit
4. Subject has two or more potential alternative approved ART drug options to consider.
5. Exclusive CCR5-tropic virus at Screening Visit
6. Plasma HIV-1 RNA < 50 copies/mL at Screening Visit
7. CD4 cell count of > 200 cells/mm3 since initiation of anti-retroviral therapy
8. CD4 cell count of > 350 cells/mm3 in preceding 24 weeks and at Screening Visit
9. Laboratory values at Screening of:

   1. Absolute neutrophil count (ANC) ≥ 750/mm3
   2. Hemoglobin (Hb) ≥ 10.5 gm/dL (male) or ≥ 9.5 gm/dL (female)
   3. Platelets ≥ 75,000 /mm3
   4. Serum alanine transaminase (SGPT/ALT) < 5 x upper limit of normal (ULN)
   5. Serum aspartate transaminase (SGOT/AST) < 5 x ULN
   6. Bilirubin (total) < 2.5 x ULN unless Gilbert's disease is present or subject is receiving atazanavir in the absence of other evidence of significant liver disease
   7. Creatinine ≤ 1.5 x ULN
10. Clinically normal resting 12-lead ECG at Screening Visit or, if abnormal, considered not clinically significant by the Principal Investigator.
11. Both male and female patients and their partners of childbearing potential must agree to use 2 medically accepted methods of contraception during the course of the study.
12. Willing and able to participate in all aspects of the study, including use of SC medication, completion of subjective evaluations, attendance at scheduled clinic visits, and compliance with all protocol requirements as evidenced by providing written informed consent.

Exclusion Criteria:

1. CXCR4-tropic virus or dual/mixed tropic (R5X4) virus determined by the Trofile™ DNA Assay
2. Hepatitis B infection as manifest by the presence of Hepatitis B surface antigen (HBsAg)
3. Any active infection or malignancy requiring acute therapy (with the exception of local cutaneous Kaposi's sarcoma)
4. Laboratory test values ≥ grade 4 DAIDS laboratory abnormality.
5. Females who are pregnant, lactating, or breastfeeding, or who plan to become pregnant during the study
6. Unexplained fever or clinically significant illness within 1 week prior to the first study dose
7. Any vaccination within 2 weeks prior to the first study dose or during the study.
8. Subjects who have failed on a maraviroc containing regimen.
9. Subjects weighing < 35kg
10. History of anaphylaxis to any oral or parenteral drugs
11. History of Bleeding Disorder or patients on anti-coagulant therapy
12. Participation in an experimental drug trial(s) within 30 days of the Screening Visit
13. Any known allergy or antibodies to the study drug or excipients
14. Treatment with any of the following:

    1. Radiation or cytotoxic chemotherapy with 30 days prior to the screening visit
    2. Immunosuppressants within 60 days prior to the screening visit
    3. Immunomodulating agents (e.g., interleukins, interferons), hydroxyurea, or foscarnet within 60 days prior to the screening visit
    4. Oral or parenteral corticosteroids within 30 days prior to the Screening Visit. Subjects on chronic steroid therapy > 5 mg/day will be excluded with the following exception:

       * Subjects on inhaled, nasal, or topical steroids will not be excluded
15. Any other clinical condition that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who remain on PRO 140 monotherapy regimen at the end of week 48 without experiencing virologic failure | 48 weeks

SECONDARY OUTCOMES:
Proportion of participants experiencing virologic failure while on PRO 140 monotherapy regimen | 48 weeks
Time to virologic failure after initiating PRO 140 monotherapy | 48 weeks
Proportion of participants achieving viral suppression (HIV-1 RNA < 50 copies/mL) after experiencing virologic failure. | 48 weeks
Time to achieving viral suppression (HIV-1 RNA < 50 copies/mL) after experiencing virologic failure | 48 weeks
Proportion of participants with viral suppression (HIV-1 RNA < 50 copies/mL) at week 48 from the start of PRO 140 Treatment Phase. | 48 weeks
Measurement of treatment adherence to the PRO 140 monotherapy regimen | 48 weeks
Total time that participants remain off combination ART regimen, defined as the time between start of PRO 140 monotherapy and restart of combination ART Regimen | 48 weeks
Mean change in CD4 cell count, at each visit within the Treatment Phase | 48 weeks
Proportion of participants experiencing emerging resistance exhibited by fold increase in maraviroc and PRO 140 FC between baseline and the time of virologic failure, as a measure of post-baseline phenotypic resistance | 48 weeks
Central Nervous System (CNS) sub-study: Level of HIV-1 RNA in CSF at T1 (prior to first dose of PRO 140), T4, T16 and VF visits | 48 weeks
Central Nervous System (CNS) sub-study: PRO 140 concentration in CSF at T1 (prior to first dose of PRO 140), T4, T16 and VF visits | 48 weeks
Central Nervous System (CNS) sub-study: Relationship between PRO 140 concentration in plasma and CSF | 48 weeks
Central Nervous System (CNS) sub-study: Relationship between PRO 140 concentration in CSF and HIV-1 RNA in CSF | 48 weeks
Genitourinary (GU) sub-study: Level of HIV-1 RNA in genital secretion at T1 (prior to first dose of PRO 140), T4, T16 and VF visits. | 48 weeks
Genitourinary (GU) sub-study: PRO 140 concentration in genital secretion at T1 (prior to first dose of PRO 140), T4, T16 and VF visits. | 48 weeks
Genitourinary (GU) sub-study: Relationship between PRO 140 concentration in plasma and genital secretion | 48 weeks
Genitourinary (GU) sub-study: Relationship between PRO 140 concentration and HIV-1 RNA in genital secretion | 48 weeks

OTHER OUTCOMES:
Tolerability of repeated subcutaneous administration of PRO 140 as assessed by study participants (using Visual Analogue Scale) | 48 weeks
Tolerability of repeated subcutaneous administration of PRO 140 as assessed by investigator evaluation of injection site reactions. | 48 weeks
Frequency of Grade 3 or 4 adverse events as defined by the DAIDS Adverse Event scale | 48 weeks
Frequency of Treatment-emergent serious adverse events | 48 weeks

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - CD03 Investigational site, La Mesa, California
  - CD03 Investigational site, Palm Springs, California
  - CD03 Investigational site, San Francisco, California
  - CD03 Investigational site, New Haven, Connecticut
  - CD03 Investigational site, Norwalk, Connecticut
  - CD03 Investigational site, Ft. Pierce, Florida
  - CD03 Investigational site, Orlando, Florida
  - CD03 Investigational site, West Palm Beach, Florida
  - CD03 Investigational site, Wichita, Kansas
  - CD03 Investigational site, Las Vegas, Nevada
  - CD03 Investigational site, New York, New York
  - CD03 Investigational site, Syracuse, New York

IPD SHARING:
Plan to Share IPD: Undecided